CLINICAL TRIAL: NCT02916368
Title: The Clinical Study of the Poorly Differentiated Head and Neck Squamous Cell
Brief Title: The Clinical Study of the Poorly Differentiated Head and Neck Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Tongren Hospital (Other)
Responsible Party: Principal Investigator, Zhigang Huang, Capital Medical University, Beijing Tongren Hospital
Other Study IDs: PDHNSCC-01609
Record Dates: First submitted 2016-09-26; First posted 2016-09-27 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- with surgery
- with chemotherapy or radiotherapy

SUMMARY:
Head and neck Squamous Cell Carcinoma (HNSCC) is one of the most common head and neck malignant tumors .Investigators found that several patients with early TNM stage and poor differentiated HNSCC had poor prognosis, yet someone with advanced TNM stage and well differentiated HNSCC had good prognosis. Hence, Investigators suggested that prognosis factors and survival rates probably related to the differentiation of HNSCC, and prognosis factor of poorly differentiated HNSCC were rare discussed and controversy. Investigating the prognostic factors of poorly differentiated HNSCC is undoubtedly crucial.

DETAILED DESCRIPTION:
Head and neck Squamous Cell Carcinoma (HNSCC) is one of the most common head and neck malignant tumors. Investigators found that several patients with early TNM stage and poor differentiated HNSCC had poor prognosis, yet someone with advanced TNM stage and well differentiated HNSCC had good prognosis. Hence, Investigators suggested that prognosis factors and survival rates probably related to the differentiation of HNSCC, and prognosis factor of poorly differentiated HNSCC were rare discussed and controversy. Investigating the prognostic factors of poorly differentiated HNSCC is undoubtedly crucial.

About this study ,inclusion criteria were the following parts:

the patients of poor differentiated HNSCC ; T1-4aN0-2M0; pathological examination: poor differentiated squamous cell carcinoma; initial treatment(primary, without surgery, radiotherapy and chemotherapy); range:18-70 years old; KPS>80; hemogram and the function of main organ such as heart, lung, liver and kidney were normal; having the endoscopy, CT and MRI before formed into different groups; sign the informed consent file, good compliance.

AND the exclusion criteria were:

uncontrollable epileptic seizure, disorder of central nervous system or unconsciousness cause by psychosis; serious and uncontrollable infection; main organ system failure (including heart ,lung ,liver and kidney); reject training; high and moderate differentiated squamous cell carcinoma

ELIGIBILITY:
Inclusion Criteria:

* Patients of poor differentiated HNSCC ;
* Patients within the stage of T1-4aN0-2M0;
* The pathological examination of the patients show poor differentiated squamous cell carcinoma;
* Patients with initial treatment(primary, without surgery, radiotherapy and chemotherapy);
* 18-70 years old;
* KPS>80;
* Hemogram and the function of main organ such as heart, lung, liver and kidney were normal
* Having the endoscopy, CT and MRI Signed the informed consent file, good compliance.

Exclusion Criteria:

* Uncontrollable epileptic seizure, disorder of central nervous system or unconsciousness cause by psychosis;
* Serious and uncontrollable infection;
* Main organ system failure (including heart ,lung ,liver and kidney); reject training;
* High and moderate differentiated squamous cell carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population were those patients with poor differentiated HNSCC from 18 to 70 years old,be in the stage of T1-4aN0-2M0 and the pathological examination shows poor differentiated squamous cell carcinoma ,also be willing take part in this study of treatment. The function of their main organ such as heart, lung, liver and kidney were normal and having the endoscopy, CT and MRI before formed into different groups.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
survival rate | 3 years

IPD SHARING:
Plan to Share IPD: Yes